CLINICAL TRIAL: NCT03502187
Title: Home-based Approaches for Subacute Low Back Pain in Active Duty: Randomized, Controlled Trial
Brief Title: Subacute Low Back Pain in Active Duty
Acronym: LBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Collaborators: Blanchfield Army Community Hospital (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HU0001-17-1-TS05 (N17-B01); 18-05885-DoD (Other: University of Tennessee)
Record Dates: First submitted 2018-03-29; First posted 2018-04-18 (Actual); Results first posted 2022-01-25 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2020-02

CONDITIONS: Subacute Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Primary Care Management (PCM) (Active Comparator): Non-specific LBP, where the cause for the pain cannot be determined, accounts for ninety percent of LBP cases.(Koes, et al, 2006) Reducing pain and continuing daily activity to prevent deconditioning are the primary therapy goals of PCM. Traditional PCM treatment of LBP will include advice/information on self-care options, over-the-counter analgesics, heat application, and remaining active.(Chou, et al., 2007; Koes, et al, 2010) Despite evidence that physical activity is effective, limiting activity remains common; individuals cite pain or re-injury fear as a limiting factor.( Lethem, et al., 1983; Poirandeau, et al., 2006; Steenstra, et al., 2016)
  Interventions: Behavioral: Primary Care Management (PCM)
- NeuromuscularElectricalStimulation(NMES) (Experimental): Rehabilitation requires activation of deep stabilizing muscle groups in the lumbopelvic region. Traditional exercises specific for these muscles are hard to teach with poor compliance. NMES is effective in stimulating these muscles, (Porcari, et al., 2005; Glaser, et al., 2001) resulting in enhanced activation, and improved performance. (Coghlan, et al., 2011) NMES devices are programmed to exercise core muscles through a series of stimulated muscle contractions. Concurrent muscle stimulation of the abdominal wall and lumbar paraspinal area has been shown to be most effective to maximally activate deep lumbar stabilizers in LBP patients. (Baek, et al., 2016) NMES provides as much pain relief as transcutaneous electric nerve stimulation (TENS) in LBP subjects. (Moore SR, Shurman J, 1997)
  Interventions: Device: NeuromuscularElectricalStimulation(NMES); Behavioral: Primary Care Management (PCM)
- Progressive Exercise Plan (PEP) (Experimental): The literature suggests that this intervention may be of benefit in military personnel with subacute LBP. (Chou, et al., 2007;Marshall PW, Murphy BA, 2006) Meta-analysis showed evidence that graded-activity exercise improved patient outcomes in subacute LBP; however, evidence for other exercise programs were inconsistent. (Hayden, et al., 2005) A strengthening program involving the trunk and abdomen muscles showed clinical reductions in low back pain and disability with high adherence. (Kendall, et al., 2015) Systematic reviews were unable to support any one type of exercise over another. The use of pain-relieving modalities combined with muscle strengthening, such as home-based electrotherapy or progressive exercise, could reduce pain and improve function more rapidly.
  Interventions: Behavioral: Progressive Exercise Plan; Behavioral: Primary Care Management (PCM)

INTERVENTIONS:
Behavioral: Progressive Exercise Plan — The goal of PEP is to reduce back pain, disability, and improve trunk flexibility, strength and endurance through controlled, gradual, progressive back exercises. PEP teaches muscle strengthening exercises and self-management strategies to promote back fitness. PEP sessions provide a standardized self-management framework for performing the exercises at home. PEP is performed every other day/week for about ~1 hour over a period of 9 weeks. PEP consists of 3 sequential phases with each phase lasting 3 weeks. Exercises become progressively more difficult and intense, focusing on back stretching and strengthening that progressively load and unload the lumbar spine by means of flexion/extension exercises. The PEP group will perform 31 exercise sessions for 60 minutes on alternating days.
  Arms: Progressive Exercise Plan (PEP)
Device: NeuromuscularElectricalStimulation(NMES) — The NMES treatment group will receive a portable battery-operated device, Recovery Back (Neurotech®, Minnetonka, MN) with a 2-garment site-specific system: back & abdomen. NMES muscle contractions will be elicited by an electrical impulse generated by the Recovery Back system. The device delivers a pre-set program of NMES using a symmetrical biphasic square pulse waveform. (Moore SR, Shurman J, 1997) The garments are light-weight, breathable fabric that wraps around the waist with precise placements for the reusable electrodes. The controller uses a rechargeable battery with charger supplied. The NMES protocol consists of 30-minutes of NMES stimulation alternating between the abdominal and lumbar site over 9-weeks (one day Back training, next day Abdominal training).
  Arms: NeuromuscularElectricalStimulation(NMES)
Behavioral: Primary Care Management (PCM) — All participants will receive standard primary care management for subacute LBP. Primary Care Management follows the clinical practice guidelines for low back pain.(Chou et al., 2007) Service members are to stay as active as possible and progressively increase their activity. Medications prescribed begin with paracetamol and NSAIDs as first-line drugs. Second-line drugs include antidepressants, benzodiazepines, tramadol, and opioids. All participants will receive an information sheet on LBP advising them to remain active and use self-care options such as heat application. To provide an attention control, the PCM only group will receive weekly communication from the study coordinator regarding pain and medication usage.

SUMMARY:
The overall objective of this project is to compare three home-managed treatment regimens for subacute low back pain: Progressive Exercise Plan (PEP), NMES (neuromuscular electrical stimulation) core strength training and standard primary care management (PCM). Each of the two treatment arms will be supplemented by Primary Care Management. The specific aim of the study is to determine whether the two treatment regimes are significantly more efficacious than standard PCM alone in improving lower back muscle strength, daily physical activity, physical function, quality of life, and symptoms associated with subacute LBP.

DETAILED DESCRIPTION:
The overall objective of this project is to compare three home-managed treatment regimens for subacute low back pain: Progressive Exercise Plan (PEP), NMES (neuromuscular electrical stimulation) core strength training and standard primary care management (PCM). The central hypothesis is that the NMES with PCM core strength training and PEP with PCM will show significantly greater improvements in muscle strength, pain, mobility/function, daily activity and quality of life (QOL) than PCM alone in military members with low back pain lasting three to eighteen weeks. The rationale for this study is that increasing torso muscle strength and decreasing pain through strength training exercises will significantly improve mobility, physical activity, QOL and reduce disability. Such outcomes could ultimately result in improved deployability, retention of military personnel and decreased economic costs in this population. The specific aims will be to determine whether the two treatment régimes are significantly more efficacious than standard PCM alone in improving lower back muscle strength, daily physical activity, physical function, quality of life, and symptoms associated with subacute LBP. After consent and baseline testing, active duty male and female subjects, ages 18 to <45, (n=135) with LBP will be randomly assigned to one of the three groups. Each of the two treatment arms will be supplemented by PCM and compared to a group receiving standard PCM alone. All groups will receive nine weeks of home therapy. Using longitudinal mixed regression models, differences in time trends for the outcome variables among controls and those in the treatment groups will be examined. In these regression analyses, the important primary measures will be expressed as a function of time, treatment group, and group-by-time interactions, while controlling for important covariates. Positive results could translate into accelerated rehabilitation, decreased symptoms and lower medical costs with better patient outcomes.

ELIGIBILITY:
Inclusion Criteria: Diagnosed with low back pain, categorized as lumbago or unspecified backache;

* greater than 3 weeks and less than 18 weeks since the onset of the episode of LBP;
* active duty military service member at the time of diagnosis;
* age ≥18 and <45 years;
* ability to provide freely given informed consent.

Exclusion Criteria:

Those who might be at risk of adverse outcomes from the study interventions will be excluded. This includes individuals with

* recurrence of LBP that is less than 3 months from prior episode;
* a significant co-morbid medical condition (such as severe hypertension, neurological disorder or pacemaker/defibrillator) in which NMES strength training or unsupervised exercise is contraindicated and would pose a safety threat or impair ability to participate;
* previous back surgeries;
* inability or unwillingness to participate in an exercise or strengthening program;
* clinical evidence of a lumbar radiculopathy;
* inability to speak and/or read English;
* pregnancy;
* vision impairment, where participant is classified as legally blind;
* unwillingness to accept random assignment; or
* a score >=23 on Center for Epidemiological Studies-Depression scale.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 133 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2020-05-28 (Actual); Study Completion 2020-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura A Talbot, PhD, EdD, RN, Principal Investigator — University of Tennessee
Locations (1):
- Blanchfield Army Community Hospital (BACH), Fort Campbell North, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koes BW, van Tulder MW, Thomas S. Diagnosis and treatment of low back pain. BMJ. 2006 Jun 17;332(7555):1430-4. doi: 10.1136/bmj.332.7555.1430. No abstract available. PMID 16777886
- [Background] Chou R, Qaseem A, Snow V, Casey D, Cross JT Jr, Shekelle P, Owens DK; Clinical Efficacy Assessment Subcommittee of the American College of Physicians; American College of Physicians; American Pain Society Low Back Pain Guidelines Panel. Diagnosis and treatment of low back pain: a joint clinical practice guideline from the American College of Physicians and the American Pain Society. Ann Intern Med. 2007 Oct 2;147(7):478-91. doi: 10.7326/0003-4819-147-7-200710020-00006. PMID 17909209
- [Background] Koes BW, van Tulder M, Lin CW, Macedo LG, McAuley J, Maher C. An updated overview of clinical guidelines for the management of non-specific low back pain in primary care. Eur Spine J. 2010 Dec;19(12):2075-94. doi: 10.1007/s00586-010-1502-y. Epub 2010 Jul 3. PMID 20602122
- [Background] Lethem J, Slade PD, Troup JD, Bentley G. Outline of a Fear-Avoidance Model of exaggerated pain perception--I. Behav Res Ther. 1983;21(4):401-8. doi: 10.1016/0005-7967(83)90009-8. No abstract available. PMID 6626110
- [Background] Poiraudeau S, Rannou F, Baron G, Henanff LA, Coudeyre E, Rozenberg S, Huas D, Martineau C, Jolivet-Landreau I, Garcia-Mace J, Revel M, Ravaud P. Fear-avoidance beliefs about back pain in patients with subacute low back pain. Pain. 2006 Oct;124(3):305-311. doi: 10.1016/j.pain.2006.04.019. Epub 2006 Jun 5. PMID 16740362
- [Background] Steenstra IA, Munhall C, Irvin E, Oranye N, Passmore S, Van Eerd D, Mahood Q, Hogg-Johnson S. Systematic Review of Prognostic Factors for Return to Work in Workers with Sub Acute and Chronic Low Back Pain. J Occup Rehabil. 2017 Sep;27(3):369-381. doi: 10.1007/s10926-016-9666-x. PMID 27647141
- [Background] Coghlan S, Crowe L, McCarthypersson U, Minogue C, Caulfield B. Neuromuscular electrical stimulation training results in enhanced activation of spinal stabilizing muscles during spinal loading and improvements in pain ratings. Annu Int Conf IEEE Eng Med Biol Soc. 2011;2011:7622-5. doi: 10.1109/IEMBS.2011.6091878. PMID 22256103
- [Background] Porcari JP, Miller J, Cornwell K, Foster C, Gibson M, McLean K, Kernozek T. The effects of neuromuscular electrical stimulation training on abdominal strength, endurance, and selected anthropometric measures. J Sports Sci Med. 2005 Mar 1;4(1):66-75. eCollection 2005 Mar 1. PMID 24431963
- [Background] Coghlan S, Crowe L, McCarthyPersson U, Minogue C, Caulfield B. Electrical muscle stimulation for deep stabilizing muscles in abdominal wall. Annu Int Conf IEEE Eng Med Biol Soc. 2008;2008:2756-9. doi: 10.1109/IEMBS.2008.4649773. PMID 19163276
- [Background] Glaser JA, Baltz MA, Nietert PJ, Bensen CV. Electrical muscle stimulation as an adjunct to exercise therapy in the treatment of nonacute low back pain: a randomized trial. J Pain. 2001 Oct;2(5):295-300. doi: 10.1054/jpai.2001.25523. PMID 14622808
- [Background] Baek SO, Cho HK, Kim SY, Jones R, Cho YW, Ahn SH. Changes in deep lumbar stabilizing muscle thickness by transcutaneous neuromuscular electrical stimulation in patients with low back pain. J Back Musculoskelet Rehabil. 2017;30(1):121-127. doi: 10.3233/BMR-160723. PMID 27341642
- [Background] Moore SR, Shurman J. Combined neuromuscular electrical stimulation and transcutaneous electrical nerve stimulation for treatment of chronic back pain: a double-blind, repeated measures comparison. Arch Phys Med Rehabil. 1997 Jan;78(1):55-60. doi: 10.1016/s0003-9993(97)90010-1. PMID 9014958
- [Background] Marshall PW, Murphy BA. Evaluation of functional and neuromuscular changes after exercise rehabilitation for low back pain using a Swiss ball: a pilot study. J Manipulative Physiol Ther. 2006 Sep;29(7):550-60. doi: 10.1016/j.jmpt.2006.06.025. PMID 16949944
- [Background] Kendall KD, Emery CA, Wiley JP, Ferber R. The effect of the addition of hip strengthening exercises to a lumbopelvic exercise programme for the treatment of non-specific low back pain: A randomized controlled trial. J Sci Med Sport. 2015 Nov;18(6):626-31. doi: 10.1016/j.jsams.2014.11.006. Epub 2014 Nov 13. PMID 25467200
- [Background] Hayden JA, van Tulder MW, Malmivaara AV, Koes BW. Meta-analysis: exercise therapy for nonspecific low back pain. Ann Intern Med. 2005 May 3;142(9):765-75. doi: 10.7326/0003-4819-142-9-200505030-00013. PMID 15867409
- [Background] Hansson TH, Bigos SJ, Wortley MK, Spengler DM. The load on the lumbar spine during isometric strength testing. Spine (Phila Pa 1976). 1984 Oct;9(7):720-4. doi: 10.1097/00007632-198410000-00012. PMID 6239393
- [Background] Ruta DA, Garratt AM, Wardlaw D, Russell IT. Developing a valid and reliable measure of health outcome for patients with low back pain. Spine (Phila Pa 1976). 1994 Sep 1;19(17):1887-96. doi: 10.1097/00007632-199409000-00004. PMID 7997920
- [Background] Fairbank JC, Couper J, Davies JB, O'Brien JP. The Oswestry low back pain disability questionnaire. Physiotherapy. 1980 Aug;66(8):271-3. No abstract available. PMID 6450426
- [Background] Revill SI, Robinson JO, Rosen M, Hogg MI. The reliability of a linear analogue for evaluating pain. Anaesthesia. 1976 Nov;31(9):1191-8. doi: 10.1111/j.1365-2044.1976.tb11971.x. PMID 1015603
- [Background] Ware JE, Jr.,, Kosinski M, Turner-Bowker DM, Gandek B. User's Manual for the SF-12v2® Health Survey with a Supplement Documenting SF-12® Health Survey. . Lincoln, RI: QualityMetric Incorporated; 2002.
- [Background] Coons SJ, Rao S, Keininger DL, Hays RD. A comparative review of generic quality-of-life instruments. Pharmacoeconomics. 2000 Jan;17(1):13-35. doi: 10.2165/00019053-200017010-00002. PMID 10747763
- [Background] Hurst NP, Ruta DA, Kind P. Comparison of the MOS short form-12 (SF12) health status questionnaire with the SF36 in patients with rheumatoid arthritis. Br J Rheumatol. 1998 Aug;37(8):862-9. doi: 10.1093/rheumatology/37.8.862. PMID 9734677
- [Background] Kantz ME, Harris WJ, Levitsky K, Ware JE Jr, Davies AR. Methods for assessing condition-specific and generic functional status outcomes after total knee replacement. Med Care. 1992 May;30(5 Suppl):MS240-52. doi: 10.1097/00005650-199205001-00024. PMID 1583936
- [Background] McHorney CA, Ware JE Jr, Lu JF, Sherbourne CD. The MOS 36-item Short-Form Health Survey (SF-36): III. Tests of data quality, scaling assumptions, and reliability across diverse patient groups. Med Care. 1994 Jan;32(1):40-66. doi: 10.1097/00005650-199401000-00004. PMID 8277801
- [Background] McHorney CA, Ware JE Jr, Raczek AE. The MOS 36-Item Short-Form Health Survey (SF-36): II. Psychometric and clinical tests of validity in measuring physical and mental health constructs. Med Care. 1993 Mar;31(3):247-63. doi: 10.1097/00005650-199303000-00006. PMID 8450681
- [Background] Chapman JR, Norvell DC, Hermsmeyer JT, Bransford RJ, DeVine J, McGirt MJ, Lee MJ. Evaluating common outcomes for measuring treatment success for chronic low back pain. Spine (Phila Pa 1976). 2011 Oct 1;36(21 Suppl):S54-68. doi: 10.1097/BRS.0b013e31822ef74d. PMID 21952190
- [Background] Marx RG, Jones EC, Allen AA, Altchek DW, O'Brien SJ, Rodeo SA, Williams RJ, Warren RF, Wickiewicz TL. Reliability, validity, and responsiveness of four knee outcome scales for athletic patients. J Bone Joint Surg Am. 2001 Oct;83(10):1459-69. doi: 10.2106/00004623-200110000-00001. PMID 11679594
- [Background] Myers JK, Weissman MM. Use of a self-report symptom scale to detect depression in a community sample. Am J Psychiatry. 1980 Sep;137(9):1081-4. doi: 10.1176/ajp.137.9.1081. PMID 7425160
- [Background] Radloff L. The CES-D scale: A self-report depression scale for research in the general population. Applied Psychological Measurement. 1977;1:385-401.
- [Background] Enright PL. The six-minute walk test. Respir Care. 2003 Aug;48(8):783-5. PMID 12890299
- [Derived] Talbot LA, Webb L, Ramirez VJ, Morrell C, Bryndziar M, Enochs K, Metter EJ. Non-pharmacological Home Therapies for Subacute Low Back Pain in Active Duty Military Personnel: A Randomized Controlled Trial. Mil Med. 2023 Jan 4;188(1-2):12-19. doi: 10.1093/milmed/usab382. PMID 34510214

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 5 participants completed the consent but withdrew from the study prior to being assigned to a group.
Groups:
- Primary Care Management (PCM): Primary Care Management (PCM): All participants received standard primary care management for subacute LBP. Primary Care Management follows the clinical practice guidelines for low back pain.(Chou et al., 2007) Service members are to stay as active as possible and progressively increase activity. Medications prescribed begin with paracetamol and NSAIDs as first-line drugs. Second-line drugs include antidepressants, benzodiazepines, tramadol, and opioids. All participants received an information sheet on LBP advising to remain active and use self-care options (e.g., heat application). To provide an attention control, the PCM only group will receive weekly communication from the study coordinator regarding pain and medication usage.
- NeuromuscularElectricalStimulation(NMES): NeuromuscularElectricalStimulation(NMES): The NMES treatment group received a portable battery-operated device, Recovery Back (Neurotech®, Minnetonka, MN) with a 2-garment site-specific system: back & abdomen. NMES muscle contractions will be elicited by an electrical impulse generated by the Recovery Back system. It delivers a pre-set program of NMES using a symmetrical biphasic square pulse waveform. (Moore SR, Shurman J, 1997) The garments are light-weight, breathable fabric wrapped around the waist with placements for reusable electrodes. The controller uses a rechargeable battery with charger supplied. The protocol consists of 30-min of NMES stimulation alternating between the abdominal and lumbar site over 9-weeks (one day Back/next day Abdominal).
  Primary Care Management (PCM): All participants received standard primary care management for subacute LBP. Primary Care Management follows the clinical practice guidelines for low back pain.(Chou et al., 2007) Service members are to stay as active as possible and progressively increase activity. Medications prescribed begin with paracetamol and NSAIDs as first-line drugs. Second-line drugs include antidepressants, benzodiazepines, tramadol, and opioids. All participants received an information sheet on LBP advising to remain active and use self-care options (e.g., heat application).
- Progressive Exercise Plan (PEP): Progressive Exercise Plan: The goal of PEP is to reduce back pain, disability, and improve trunk flexibility, strength and endurance through controlled, gradual, progressive back exercises. PEP teaches muscle strengthening exercises and self-management strategies to promote back fitness. PEP sessions provide a standardized self-management framework for performing the exercises at home. PEP is performed every other day/week for about ~1 hour over a period of 9 weeks. PEP consists of 3 sequential phases with each phase lasting 3 weeks. Exercises become progressively more difficult and intense, focusing on back stretching and strengthening that progressively load and unload the lumbar spine by means of flexion/extension exercises. The PEP group will perform 31 exercise sessions for 60 minutes on alternating days.
  Primary Care Management (PCM): All participants received standard primary care management for subacute LBP. Primary Care Management follows the clinical practice guidelines for low back pain.(Chou et al., 2007) Service members are to stay as active as possible and progressively increase activity. Medications prescribed begin with paracetamol and NSAIDs as first-line drugs. Second-line drugs include antidepressants, benzodiazepines, tramadol, and opioids. All participants received an information sheet on LBP advising to remain active and use self-care options (e.g., heat application).
Period: Overall Study
Arm/Group | Primary Care Management (PCM) | NeuromuscularElectricalStimulation(NMES) | Progressive Exercise Plan (PEP)
Started | 43 | 43 | 42
Completed | 34 | 36 | 34
Not Completed | 9 | 7 | 8
Not completed — Withdrawal by Subject | 4 | 3 | 3
Not completed — Lost to Follow-up | 5 | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Primary Care Management (PCM) | NeuromuscularElectricalStimulation(NMES) | Progressive Exercise Plan (PEP) | Total
Number analyzed (Participants) | 43 | 43 | 42 | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.84 (5.66) | 25.47 (5.22) | 25.05 (5.47) | 25.5 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 7 | 22
  Male | 35 | 36 | 35 | 106
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 24 | 24 | 24 | 72
  African American | 12 | 13 | 12 | 37
  Asian/Pacific | 3 | 2 | 1 | 6
  Amer. Indian/Alaska Native | 1 | 1 | 0 | 2
  Multi-racial | 3 | 3 | 5 | 11
Mechanism of Injury [Count of Participants; unit: Participants]
  Sports | 0 | 2 | 1 | 3
  Work | 9 | 6 | 11 | 26
  Military Training | 27 | 28 | 24 | 79
  Other | 7 | 7 | 6 | 20
Rank [Count of Participants; unit: Participants]
  Enlisted | 39 | 40 | 42 | 121
  Warrant Officer | 0 | 2 | 0 | 2
  Officer | 4 | 1 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Lower Back Strength-Extension
Description: Torso extension muscle strength is measured with a modified version of the U of Michigan strength test system (Workability Systems, West Chester, Ohio) and a Chattanooga-Baseline® Hand Dynamometer - Digital LCD Gauge - ER™ 300 lb capacity (DJO Global, Chattanooga, Vista, CA USA). To measure trunk extension, the participant stands with their lower anterior abdomen against the padded board. The belt is placed around the posterior back and under the arms. Participants pull against the belt as forcefully as possible. Participants perform two maximal efforts maintaining each voluntary isometric exertion for 5 seconds, separated by 30-second rest; the highest value of the two trials will be accepted.
Time Frame: 0, 3, 6, and 9 weeks
Measure: Mean (Standard Deviation); unit: kg-Force
Arm/Group | Primary Care Management (PCM) | NeuromuscularElectricalStimulation(NMES) | Progressive Exercise Plan (PEP)
Number analyzed (Participants) | 43 | 43 | 42
kg-Force
  Week 0 | 54.5 (28.9) | 50.2 (25.4) | 49.2 (27.2)
  Week 3 | 57.5 (33.1) | 61.4 (34.6) | 54.6 (31.0)
  Week 6 | 68.2 (36.9) | 69.0 (33.4) | 53.1 (30.1)
  Week 9 | 69.4 (30.7) | 69.3 (39.3) | 55.1 (23.6)

2. Primary Outcome: Lower Back Strength-Flexion
Description: Torso flexion muscle strength is measured with a modified version of the U of Michigan strength test system (Workability Systems, West Chester, Ohio) and a Chattanooga-Baseline® Hand Dynamometer - Digital LCD Gauge - ER™ 300 lb capacity (DJO Global, Chattanooga, Vista, CA USA). For trunk flexion, the participant stands in the apparatus, buttocks against the padded board, the superior edge level with the iliac crest. A canvas belt is around the chest and under the arms horizontal to the force-measuring dynamometer on the apparatus frame. Participants pull against the belt as forcefully as possible. Participants perform two maximal efforts maintaining each voluntary isometric exertion for 5 seconds, separated by 30-second rest; the highest value of the two trials will be accepted.
Time Frame: 0, 3, 6, and 9 weeks
Measure: Mean (Standard Deviation); unit: kg-Force
Arm/Group | Primary Care Management (PCM) | NeuromuscularElectricalStimulation(NMES) | Progressive Exercise Plan (PEP)
Number analyzed (Participants) | 43 | 43 | 42
kg-Force
  Week 0 | 51.6 (29.7) | 48.8 (27.7) | 43.7 (23.1)
  Week 3 | 52.1 (29.6) | 57.9 (30.5) | 47.7 (26.3)
  Week 6 | 65.6 (39.9) | 63.7 (29.6) | 44.4 (26.3)
  Week 9 | 65.1 (29.9) | 60.9 (30.9) | 47.9 (22.5)

3. Secondary Outcome: Current Pain Severity
Description: The Visual Analog Scale (VAS) of pain will be used to assess pain at rest and after activity. (Revill et al., 1976) Participants will complete this scale following the push-ups, sit-ups, 6-minute walk and the lumbar trunk muscle test. This VAS pain subscale is a 10-cm horizontal line index with descriptive anchors at each end. At the far left (0.0 cm) is "no pain" and at the far right (10 cm) is "worst possible pain". The participant is instructed to place a vertical line at some point between the anchors to describe their level of pain.
Time Frame: 0, 3, 6, 9 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Primary Care Management (PCM) | NeuromuscularElectricalStimulation(NMES) | Progressive Exercise Plan (PEP)
Number analyzed (Participants) | 43 | 43 | 42
score on a scale
  Week 0 | 4.43 (2.0) | 4.57 (2.2) | 4.78 (2.0)
  Week 3 | 3.88 (2.6) | 4.54 (2.3) | 4.47 (2.2)
  Week 6 | 4.03 (2.5) | 3.96 (2.9) | 4.70 (2.6)
  Week 9 | 3.28 (2.6) | 4.07 (3.1) | 3.93 (2.7)

4. Secondary Outcome: Impact of Bodily Pain on Normal Work Measured by SF12v2
Description: The Short Form Health Survey Version 2.0 (SF-12v2) Health Survey will be used to determine each participant's overall impact of bodily pain on normal work. The SF12v2 has a question that asks participants to assess the impact of pain on normal work during the previous 4 weeks using options ranging from Not at all to Extremely. Responses are translated to numerical scores ranging from 0 to 100. Higher scores indicate less impact of bodily pain.
Time Frame: 0, 3, 6, 9 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Primary Care Management (PCM) | NeuromuscularElectricalStimulation(NMES) | Progressive Exercise Plan (PEP)
Number analyzed (Participants) | 43 | 43 | 42
score on a scale
  Week 0 | 53.6 (22.5) | 44 (27.5) | 47.6 (19.0)
  Week 3 | 59.0 (24.0) | 58.8 (22.2) | 55.9 (22.2)
  Week 6 | 59.2 (23.2) | 61.4 (26.6) | 58.6 (25.1)
  Week 9 | 72.0 (23.2) | 72.1 (21.1) | 65.8 (23.2)

5. Secondary Outcome: Physical Activity
Description: Physical activity will be measured using the Fitbit Charge 2 (San Francisco, CA). The Charge 2 is a wrist-worn three-axis accelerometer that measures steps walked, distance traveled, energy expenditure and floors climbed. The unique feature of this device is a wireless function that automatically uploads data to designated mobile phone devices or computers. Physical Activity is reported as average Kcal expended during a seven day period.
Time Frame: 0, 3, 6, 9 Weeks
Measure: Mean (Standard Deviation); unit: Kcal
Arm/Group | Primary Care Management (PCM) | NeuromuscularElectricalStimulation(NMES) | Progressive Exercise Plan (PEP)
Number analyzed (Participants) | 43 | 43 | 42
Kcal
  Week 0 | 2733 (1024) | 3005 (932) | 2912 (1019)
  Week 3 | 2691 (955) | 2950 (854) | 2809 (1040)
  Week 6 | 2599 (843) | 2955 (942) | 2609 (934)
  Week 9 | 2605 (942) | 2922 (1107) | 2559 (700)

6. Secondary Outcome: Mobility/Function Measured by the 2-minute Push-up Test
Description: The 2-minute push-up test evaluates upper body endurance and strength as well as the stabilizing torso muscles of the abdomen and back. Starting in a prone position, the participant is positioned with their hands on the ground (shoulder width apart), toes in contact with the floor, spine parallel to the floor, elbows and hips in extension. The body moves as a single rigid unit and is lowered to the ground until elbows are at 90° angle. The body is then returned to the starting position by pushing the arms up to full extension. A push-up is counted if the elbows were brought to flexion of 90° or greater and then return to full extension, while keeping the body elevated on the toes. The number of push-ups performed in 2-minutes is recorded.
Time Frame: 0, 3, 6, 9 Weeks
Measure: Mean (Standard Deviation); unit: Number of push-ups
Arm/Group | Primary Care Management (PCM) | NeuromuscularElectricalStimulation(NMES) | Progressive Exercise Plan (PEP)
Number analyzed (Participants) | 43 | 43 | 42
Number of push-ups
  Week 0 | 46.9 (14.4) | 41.1 (18.2) | 43.7 (18.4)
  Week 3 | 46.0 (16.3) | 40.3 (20.4) | 47.4 (16.8)
  Week 6 | 45.9 (14.6) | 42.3 (18.7) | 42.2 (18.7)
  Week 9 | 46.2 (18.1) | 46.0 (22.9) | 46.3 (17.2)

7. Secondary Outcome: Mobility/Function Measured by the 2-minute Sit-up Test
Description: The 2-minute sit-up test measures trunk flexion and abdominal endurance. Starting in a supine position, the knee joints are flexed at a 90° angle, with fingers behind the head, soles of the feet and shoulder blades in contact with the floor. With the command to begin, the upper body is raised forward by flexing the abdominal muscles and then lowered. A sit-up is counted if the hands are behind the head, bringing the base of the spine to a vertical position and then returning the shoulder blades to the floor. The number of repetitions performed in 2 minutes is recorded.
Time Frame: 0, 3, 6, 9 Weeks
Measure: Mean (Standard Deviation); unit: Number of sit-ups
Arm/Group | Primary Care Management (PCM) | NeuromuscularElectricalStimulation(NMES) | Progressive Exercise Plan (PEP)
Number analyzed (Participants) | 43 | 43 | 42
Number of sit-ups
  Week 0 | 44.4 (17.6) | 35.5 (21.4) | 41.5 (15.2)
  Week 3 | 44.9 (18.8) | 38.7 (21.5) | 43.2 (15.3)
  Week 6 | 45.6 (18.4) | 43.2 (15.2) | 40.8 (14.9)
  Week 9 | 51.0 (14.5) | 43.5 (18.2) | 45.0 (13.0)

8. Secondary Outcome: Mobility/Function Measured by the 6-minute Walk Test
Description: The 6-Minute Walk Test (6-MWT) measures the distance a participant walks at a "fast" pace over a 6-minute period. Participants will "walk as quickly as you can" with the opportunity to stop and rest if required. This test measures functional capacity of walking. Healthy adults are expected to walk between 400 and 700 meters [1300-2300 feet] on the 6-minute walk test (Enright, 2003). Outcomes are reported in feet walked.
Time Frame: 0, 3, 6, 9 Weeks
Measure: Mean (Standard Deviation); unit: Number of feet
Arm/Group | Primary Care Management (PCM) | NeuromuscularElectricalStimulation(NMES) | Progressive Exercise Plan (PEP)
Number analyzed (Participants) | 43 | 43 | 42
Number of feet
  Week 0 | 1940 (253) | 1868 (335) | 1858 (225)
  Week 3 | 2020 (245) | 1889 (320) | 1882 (235)
  Week 6 | 1996 (280) | 1925 (237) | 1904 (257)
  Week 9 | 2041 (271) | 1883 (427) | 1924 (283)

9. Secondary Outcome: Depressive Symptoms-Center for Epidemiologic Studies Depression (CES-D) Scale
Description: The Center for Epidemiologic Studies Depression (CES-D) scale is a self-report questionnaire that contains 20 items. Participants were asked to rate how often over the past week they experienced symptoms associated with depression. Scores range from 0-60 with high scores denoting greater depressive symptoms. CES-D scores were recorded at baseline (0 weeks) and subsequent visits. If the baseline score was greater than 23 the participants were not randomized.
Time Frame: 0, 3, 6, 9 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Primary Care Management (PCM) | NeuromuscularElectricalStimulation(NMES) | Progressive Exercise Plan (PEP)
Number analyzed (Participants) | 43 | 43 | 42
score on a scale
  Week 0 | 6.84 (6.29) | 6.05 (6.07) | 6.26 (5.50)
  Week 3 | 7.78 (6.10) | 6.46 (4.72) | 7.12 (7.25)
  Week 6 | 6.13 (6.31) | 6.55 (6.40) | 8.06 (6.96)
  Week 9 | 5.70 (6.11) | 6.20 (7.28) | 7.63 (7.25)

ADVERSE EVENTS:
Time Frame: 9 weeks
Arm/Group | Primary Care Management (PCM) | NeuromuscularElectricalStimulation(NMES) | Progressive Exercise Plan (PEP)
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/43 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/43 | 0/42
Other Adverse Events (participants affected / at risk) | 0/43 | 0/43 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-04-17): https://cdn.clinicaltrials.gov/large-docs/87/NCT03502187/Prot_002.pdf
  • Statistical Analysis Plan (2018-04-17): https://cdn.clinicaltrials.gov/large-docs/87/NCT03502187/SAP_003.pdf
  • Informed Consent Form (2020-01-08): https://cdn.clinicaltrials.gov/large-docs/87/NCT03502187/ICF_001.pdf